CLINICAL TRIAL: NCT05114317
Title: Pain Characteristics, Intensity, Patterns, Impact and Quality of Life in Women With Lipoedema: an Online Survey
Brief Title: Characteristics of Pain in Women With Lipoedema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Other Study IDs: EC2_CWT
Record Dates: First submitted 2021-06-02; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Lipedema
Keywords: Pain; Emotional status; Quality of life
MeSH Terms: conditions — Lipedema; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Lipoedema: No interventions administered.

SUMMARY:
This observational study will seek to investigate the following questions in women with lipoedema:

* pain characteristics, intensity and patterns of pain
* the relationships between the characteristics, intensity and patterns of pain and age, ethnicity, location, employment status, levels of anxiety/depression, walking ability, ability to work, relations with other people, impact on sleep and quality of life.
* the impact of pain treatments or medications on the intensity of pain. The information will be collected via an online survey and participants will be recruited through social media platforms.

DETAILED DESCRIPTION:
Lipoedema is a chronic adipose tissue disorder that occurs almost exclusively in women and affects approximately 11% worldwide. Pain is a recurring feature described by people with lipoedema (pwL) with a recent study reporting 88.3% of patients indicating pain as a clinical feature. It has been suggested, with chronic long-term conditions, that the pain people experience can be moulded by a myriad of elements.This includes biomedical, psychosocial (e.g. patients' beliefs, expectations, and mood), and behavioural factors (e.g. context, responses by significant others). PwL often experience significant impairment in their daily activities and quality of life. It has further been found that psychological and the biomedical consequences of lipoedema can increase the chances of anxiety and depression which can subsequently further impact on quality of life and pain experience.

This observational study will seek to investigate the following questions in women with lipoedema:

* pain characteristics, intensity and patterns of pain
* the relationships between the characteristics, intensity and patterns of pain and age, ethnicity, location, employment status, levels of anxiety/depression, walking ability, ability to work, relations with other people, impact on sleep and quality of life.
* the impact of pain treatments or medications on the intensity of pain. INformation about pain characteristics, demographics, mood, functional ability and quality of life will be collected via an online survey and participants will be recruited through social media platforms.

ELIGIBILITY:
Inclusion Criteria:

* Women with lipoedema
* 16 years and older

Exclusion Criteria:

- Inability to provide consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Study Population: Women with lipoedema.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - short form | Only once at participation, the study duration is approximately 2 years
  The Brief Pain Inventory - Short Form is a simple, 9 question self-reporting tool that expands on other questionnaires such as the McGill pain questionnaire which focuses more on the quality of pain. The questionnaire allows the individual to rate the severity of pain and it also looks at how pain affects daily functions and discloses the site of pain in the past 24 hours. Within the questionnaire there are four severity questions looking at pain 'at least', 'at worst' (both in the last 24 hours), 'on average' and 'now' using a Likert scale with 0 = no pain to 10 = pain as bad as you can imagine. Seven pain interference domains are also included in the questionnaire covering general activity, mood, walking ability, normal work, relations with others, sleep and enjoyment of life. These are also measured on a Likert scale with 0 = no interference to 10 = interferes completely.

SECONDARY OUTCOMES:
Symptoms severity scale | During study, only once at participation - 2 years
  Symptom severity will be recorded using a 5 - point Likert scale with 1 = no problem to 5 = extremely severe. These symptoms include:
  1. swelling of the affected areas,
  2. loose connective tissues around the knee joints,
  3. tenderness,
  4. easy or spontaneous bruising, and
  5. presence of spider veins.
Depression, Anxiety and Stress Scale - 21 | Only once at participation, the study duration is approximately 2 years
  The Depression, Anxiety and Stress Scale - 21 is a a self-reporting questionnaire with three scales measuring three negative emotional states: depression, anxiety, and stress. Within the questionnaire, each of the three scales contain 7 items with the scores of these items totalled. Each item is score on a likert scale of 0 to 3: 0 being ' did not apply to me at all', 1 being 'applied to me to some degree, or some of the time, 2 being 'applied to me to a considerable degree' or a good part of the time', 3 being 'applied to me very much or most of the time'.
World Health Organization Quality of Life Assessment | Only once at participation, the study duration is approximately 2 years
  The World Health Organization Quality of Life Assessment is a shorter version of the initially developed questionnaire with 100 items, with this shorter version containing 26 items. It measures the broad domains of physical health, psychological health, social relationships, and environment. For each of these domains a mean score is produced for use within research and analysis. The items are rated on a 5-point Likert scale (low score of 1to high score of 5) to determine the raw item score. The the mean for each domain is calculated. After which, the domain score is multiplied by 45 to transform the domain score into a scaled score. A high score indicates a higher quality of life.

OTHER OUTCOMES:
Demographic questionnaire | Only once at participation, the study duration is approximately 2 years
  Data for the following variables will be collected from the participants:
  * age
  * ethnicity
  * country of domicile
  * employment status
  * height
  * weight
  * number of comorbidities
  * walking aid usage
  * time of awareness of lipoedema
  * type of lipoedema

CONTACTS AND LOCATIONS:
Overall Officials: Chee Wee Tan, PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom